CLINICAL TRIAL: NCT07252661
Title: An Open-Label, Phase 1 Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of ACC-1898 (Tyrosine Kinase Inhibitor) in Adult Participants With Advanced Solid Tumors.
Brief Title: Study of ACC-1898 in Adult Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AccSalus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACC-1898-101
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Renal Cell Carcinoma; Thyroid Carcinoma, Medullary; Thyroid Carcinoma Primary Differentiated; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Melanoma; Gall Bladder Cancer; Advanced Solid Tumor
Keywords: Advanced Solid Tumors; Metastatic Cancer; Tyrosine Kinase Inhibitor; VEGFR; MET; RET; AXL; Multi-target TKI; ACC-1898
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Thyroid cancer, medullary; Melanoma; Gallbladder Neoplasms; Neoplasm Metastasis | interventions — 3-(3'-adamantan-1-yl-4'-methoxybiphenyl-4-yl)-2-propenoic acid

STUDY DESIGN:
Intervention Model Description: Open-label, dose-escalation study followed by expansion at the recommended dose in participants with advanced solid tumors.
Masking Description: This is an open-label study; no masking or blinding procedures are applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receive ACC-1898 tablets orally once daily (QD) in 21-day cycles (Experimental): Dose-Escalation (Part 1): Determine the maximum tolerated dose (MTD) and/or optimal biologic dose (OBD) using an Accelerated Titration → Bayesian Optimal Interval (ATD-BOIN) design.
  Treatment continues until disease progression, unacceptable toxicity, withdrawal, or study completion
  Interventions: Drug: ACC-1898
- ACC-1898 Dose Expansion Cohorts (Experimental): Participants will receive ACC-1898 tablets orally once daily (QD) in repeating 21-day cycles at dose levels determined from Part 1 (dose escalation).
  This Phase 1b dose-expansion phase will enroll patients with selected advanced or metastatic solid tumors to further characterize the safety, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of ACC-1898 at the recommended Part 2 dose(s).
  Up to three tumor-specific expansion cohorts may be opened. Within each indication, participants may be randomized between two ACC-1898 dose levels that demonstrated acceptable safety and evidence of activity in Part 1.
  Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or study completion.
  Paired tumor biopsies and optional blood samples will be collected to explore biomarker and PK/PD correlations.
  Interventions: Drug: ACC-1898

INTERVENTIONS:
Drug: ACC-1898 — ACC-1898 is an oral small-molecule tyrosine kinase inhibitor (TKI).
  Administered once daily by mouth in continuous 21-day cycles.
  Starting doses range from 80 mg to 300 mg QD, with possible intra-patient dose modifications.
  Arm(s)/Group(s):
  * Arm 1 - ACC-1898 Monotherapy
  * Arm 2 - ACC-1898 Monotherapy
  Route of Administration:
  Oral (tablet)
  Dose Form:
  Film-coated tablet (20 mg and 40 mg strengths)
  Treatment Duration:
  Up to 2 years or until disease progression or unacceptable toxicity.
  Other Names: ST-1898

SUMMARY:
This is a research study of an experimental drug called ACC-1898. ACC-1898 is an oral tyrosine kinase inhibitor (TKI) that blocks several proteins kinases which may help cancer cells grow and spread.

The purpose of this Phase 1 clinical trial is to find a safe dose of ACC-1898 and to understand how the body absorbs, distributes, and eliminates the drug (pharmacokinetics / PK). The study will also look for early signs that ACC-1898 may slow or shrink tumors and explore possible biological markers related to drug activity.

Adults with advanced or metastatic solid tumors who have no remaining standard treatment options may take part.

All participants will receive ACC-1898 tablets by mouth once daily in repeating 21-day cycles. Treatment may continue for up to two years if the cancer does not worsen and side effects are manageable.

Safety information, laboratory results and imaging scans (CT or MRI) will be collected regularly.

The study will first test different dose levels (dose-escalation phase) and may later expand enrollment in selected tumor types once a recommended dose is found.

DETAILED DESCRIPTION:
Study Design:

ACC-1898-101 is an open-label, multicenter, interventional Phase 1 study sponsored by AccSalus Biosciences Inc. (IND #177222). The trial evaluates the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of ACC-1898 in adults with advanced solid tumors that are unresponsive to or ineligible for standard therapies.

Rationale:

Aberrant activation of receptor tyrosine kinases (RTKs) drives tumor proliferation, angiogenesis, and resistance to therapy.

ACC-1898 (also known as ST-1898) is a small-molecule inhibitor designed to block several RTK pathways simultaneously. Nonclinical studies demonstrated broad antitumor activity and favorable oral bioavailability, while early clinical experience (≈ 100 patients in prior Asian trials) showed a manageable safety profile with preliminary efficacy.

Objectives:

Primary - determine the maximum tolerated dose (MTD) and/or optimal biologic dose (OBD) and characterize safety.

Secondary - define PK parameters (Cmax, AUC, t½, CL/F, Vz/F) after single and repeated dosing.

AUC: Area Under the Plasma Concentration-Time Curve t½: Terminal Elimination Half-Life CL/F: Apparent Oral Clearance Vz/F: Apparent Volume of Distribution

Exploratory - evaluate objective response rate (ORR), disease control rate (DCR), duration of response (DOR), progression-free survival (PFS), and biomarker or PK/PD correlations.

Methods:

Approximately 40 participants will be enrolled during the dose-escalation part (Part 1) using an Accelerated Titration → Bayesian Optimal Interval (ATD (Accelerated Titration Design) -BOIN) design with planned dose levels of 80-300 mg once daily.

Treatment continues in 21-day cycles until disease progression, unacceptable toxicity, withdrawal, or study completion.

After identification of an MTD or recommended Part 2 dose, expansion cohorts may be opened for selected tumor types

Assessments:

Safety evaluations include adverse events (AEs), clinical laboratory tests, vital signs and imaging per RECIST (Response Evaluation Criteria in Solid Tumors) 1.1.

PK sampling occurs intensively on Cycle 1 Day 1 and 15 and at steady-state in subsequent cycles.

Duration:

Each participant's involvement includes up to 28 days for screening, treatment for up to 2 years, and safety follow-up approximately 28 days after the last dose.

Data Oversight:

A Cohort Review Committee (CRC) serves as the data-monitoring body to review emerging safety and PK data before escalation or expansion decisions.

Benefit-Risk Consideration:

For patients with no remaining standard therapy, ACC-1898 offers a rational mechanism to target multiple oncogenic RTKs in a single oral agent. Known class-related risks are proactively managed through eligibility criteria, close monitoring, and prespecified dose-modification rules.

ELIGIBILITY:
Inclusion Criteria (highlights):

Adults (≥ 18 years) with histologically confirmed advanced or metastatic solid tumors that have progressed after standard therapy or for which no effective standard option exists.

At least one measurable lesion per RECIST v1.1.

ECOG (Eastern Cooperative Oncology Group) Performance Status 0-1 (2 may be allowed with Medical Monitor approval).

Resolved acute effects from prior therapy to ≤ Grade 1 per CTCAE v5.0.

Adequate organ function (hematologic, hepatic, renal).

Able to swallow oral medication and comply with study requirements.

Signed informed consent.

Women of childbearing potential must have a negative pregnancy test and use highly effective contraception during and for 180 days after treatment; men must use condoms and avoid sperm donation for 120 days post-treatment.

Exclusion Criteria (highlights):

Known primary CNS (central nervous system) malignancy or symptomatic brain metastases requiring supraphysiologic steroids (unless stable ≥ 3 months after therapy).

Active or uncontrolled infection (including HBV, HCV, HIV) not meeting protocol control criteria.

HBV: Hepatitis B Virus HCV: Hepatitis C Virus HIV: Human Immunodeficiency Virus

Significant GI disease that could impair oral drug absorption (e.g., unresolved Grade > 1 nausea/diarrhea).

Active liver or biliary disease (except stable metastases or Gilbert's syndrome).

Baseline QTcF (QT Interval Corrected Using Fridericia Formula) > 450 msec (men) or > 470 msec (women), clinically significant ECG abnormalities, or heart rate < 45 bpm unless approved by cardiology review.

Pregnant or breastfeeding women.

Any other medical condition that, in the investigator's judgment, would interfere with study participation or pose unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) Part 1 (Dose Escalation) | Cycle 1 (each cycle = 21 days)
  Occurrence of DLTs within the first treatment cycle to determine the maximum tolerated dose (MTD) and/or recommended Part 2 dose (OBD).
Treatment-Emergent Adverse Events (TEAEs) | From first dose through 28 days after last dose (up to 2 years)
  Incidence, severity, and relationship of TEAEs graded per CTCAE v5.0.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) Part 1 (Pharmacokinetics) | Cycle 1 Day 1 and Day 15 (Cycle length = 21 days)
  Maximum plasma concentration after oral dosing, derived from individual plasma concentration-time profiles.
Area Under the Concentration-Time Curve (AUC₀-last) Part 1 (Pharmacokinetics) | Cycle 1 Day 1 and Day 15 (Cycle length = 21 days)
  Total drug exposure from dosing to last measurable concentration.
AUC₀-τ (steady-state interval) Part 1 (Pharmacokinetics) | Cycle 1 Day 15 (Cycle length = 21 days)
  Exposure during one 24-hour dosing interval at steady state
AUC₀-∞ Part 1 (Pharmacokinetics) | Cycle 1 Day 1 (Cycle length = 21 days)
  Total systemic exposure extrapolated to infinity after a single dose.
Terminal Half-Life (t½) Part 1 (Pharmacokinetics) | Cycle 1 Day 1 and Day 15 (Cycle length = 21 days)
  Time for plasma concentration to decrease by 50 % during terminal phase.
Apparent Oral Clearance (CL/F) Part 1 (Pharmacokinetics) | Cycle 1 Day 15 (Cycle length = 21 days)
  Dose/AUC representing systemic clearance after oral dosing.
Apparent Volume of Distribution (Vz/F) Part 1 (Pharmacokinetics) | Cycle 1 Day 15 (Cycle length = 21 days)
  Extent of drug distribution following oral administration.
Minimum Observed Plasma Concentration (Cmin) Part 1 (Pharmacokinetics) | Cycle 1 Day 15 (Cycle length = 21 days)
  Trough plasma level within dosing interval at steady state.
Accumulation Ratio for AUC (AR-AUC) Part 1 (Pharmacokinetics) | Cycle 1 Day 15 vs Day 1 (Cycle length = 21 days)
  Ratio of AUC after repeated versus single dosing.
Accumulation Ratio for Cmax (AR-Cmax) Part 1 (Pharmacokinetics) | Cycle 1 Day 15 vs Day 1 (Cycle length = 21 days)
  Ratio of Cmax after repeated versus single dosing.

IPD SHARING:
Plan to Share IPD: No
This early-phase, first-in-human study is designed primarily to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of ACC-1898.
  Individual participant data (IPD) will not be shared publicly because the dataset may contain information that could compromise participant privacy or study integrity and is not suitable for broader distribution at this stage of development.
  Aggregate summaries of safety and pharmacokinetic results may be provided in future scientific publications or regulatory submissions.